CLINICAL TRIAL: NCT00231166
Title: A Phase I, Dose-finding Trial of HCD122, an Anti-CD40 Monoclonal Antibody, in Patients With Multiple Myeloma That is Relapsed or Has Not Responded to Prior Therapy (CHIR1212-C12101)
Brief Title: Safety, Efficacy, Dose-finding Study of a Monoclonal Antibody in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHCD122A2102; NCT00304109 (obsolete NCT alias)
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Multiple Myeloma
Keywords: dose-finding; monoclonal antibody; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — lucatumumab

ARMS (1):
- HCD122 (Experimental)
  Interventions: Drug: HCD122

INTERVENTIONS:
Drug: HCD122

SUMMARY:
The purpose of this study is to determine the highest tolerated dose, safety and activity of HCD122 in patients with Multiple Myeloma who are relapsed after receiving prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of MM requiring treatment
* Refractory or Relapsed Disease
* At least one prior treatment regimen
* Male or Female
* >18 years of age

Exclusion Criteria:

* Prior Allogeneic bone marrow transplant (prior autologous transplant allowed)
* Intracranial disease or epidural disease
* Clinically significant cardiac dysfunction or other significant organ dysfunction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety, pharmacokinetics and pharmacodynamics at multiple doses | At the completion of each dose escalation cohort

SECONDARY OUTCOMES:
Clinical response after various doses | Once a month

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (7):
- United States (5):
  - Dana Farber Cancer Institute StudyCoordinator:CHCD122A2102, Boston, Massachusetts
  - St. Vincent's Comprehensive Cancer Center Dept. of St. Vincent's Cancer, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania--Abramson Cancer Center StudyCoordinator:CHCD122A2102, Philadelphia, Pennsylvania
  - Fred Hutchinson Cancer Research Center Dept. of FHCRC, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Prahran, Victoria